CLINICAL TRIAL: NCT00437372
Title: A Phase IB, Open-Label, Safety Study of the Combination of Sunitinib and Radiation for the Treatment of Patients With Cancer
Brief Title: Phase IB Study Using Sunitinib Plus Radiation Therapy for Cancer Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sidney Kimmel Cancer Center at Thomas Jefferson University (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Organization: Thomas Jefferson University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06C.549; 2006-30 (Other: CCRRC); JT 1208 (Other: JeffTrial Number)
Record Dates: First submitted 2007-02-20; First posted 2007-02-21 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Cancer; Head and Neck Cancer; Pelvic Cancer; Nervous System Neoplasms; Thoracic Neoplasms
Keywords: solid tumor; central nervous system; head and neck; thorax; pelvic area
MeSH Terms: conditions — Neoplasms; Head and Neck Neoplasms; Pelvic Neoplasms; Nervous System Neoplasms; Thoracic Neoplasms | interventions — Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Sunitinib plus Radiation (Experimental): Sunitinib plus Radiation
  Interventions: Drug: Sunitinib; Radiation: External Beam Radiation Therapy

INTERVENTIONS:
Drug: Sunitinib — The use of the FDA approved drug sunitinib, used in an "off-label" manner with external beam radiation therapy.
  Other Names: Sutent; SU11248
Radiation: External Beam Radiation Therapy — Radiotherapy will be administered Monday through Friday for a maximum of 8 weeks. Total dose will depend on the patient's disease site.
  Other Names: External Beam Radiotherapy; Teletherapy

SUMMARY:
This study is using the combination of radiation and antiangiogenic agents (agents that destroy existing blood vessels) seems to be an approach to tumor cure.

DETAILED DESCRIPTION:
The combination of ionizing radiation and antiangiogenic agents seems to be a counterintuitive approach to tumor cure because oxygen is a potent radiosensitizer and a reduction in oxygen concentration would be expected following a reduction in tumor vasculature after antiangiogenic treatment.

ELIGIBILITY:
Inclusion Criteria:

* Minimum 2 week course of radiation therapy
* Solid tumors of the central nervous system, head and neck, thorax, and pelvis

Exclusion Criteria:

* Major surgery or radiation therapy within 4 weeks starting study treatment
* Grade 3 hemorrhage within 4 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2007-03; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the safety and toxicity profile of sunitinib when used with concurrent radiation therapy | 2 years
  The purpose of this study is to determine the safety of the combination of the antiangiogenic, sunitinib, when combined with external beam radiotherapy.

SECONDARY OUTCOMES:
To measure urine VEGF | 2 years
  Urine VEGF may be a biomarker of response. This translational approach may be useful to determine who benefits from treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Adam P Dicker, MD, PhD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University, Philadelphia, Pennsylvania, United States

REFERENCES:
- See also: Kimmel Cancer Center at Thomas Jefferson University, an NCI-Designated Cancer Center — http://www.KimmelCancerCenter.org
- See also: Thomas Jefferson University Hospitals — http://www.JeffersonHospital.org